CLINICAL TRIAL: NCT01909115
Title: Randomized Trial of Two Maintenance Doses of Vitamin D and Trace Element Status in Children With Chronic Kidney Disease
Brief Title: Two Vitamin D Dosing Strategies in Children With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Larry Greenbaum, MD, PhD, Professor of Pediatric Nephrology and Division Director of Pediatric Nephrology, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00067067; EmoryPedNeph-001 (Other: Other)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1000 IU of Vitamin D Daily (Active Comparator): Participants randomized to take a 1000 IU capsule of Vitamin D every day for 6 months.
  Interventions: Drug: 1000 IU of Vitamin D3
- 4000 IU of Vitamin D Daily (Experimental): Participants randomized to take a 4000 IU capsule of Vitamin D capsule every day for 6 months.
  Interventions: Drug: 4000 IU of Vitamin D3

INTERVENTIONS:
Drug: 1000 IU of Vitamin D3 — 1000 IU of Vitamin D will be administered in capsule form, once daily.
  Arms: 1000 IU of Vitamin D Daily
Drug: 4000 IU of Vitamin D3 — 4000 IU of Vitamin D will be administered in capsule form, once daily.
  Arms: 4000 IU of Vitamin D Daily

SUMMARY:
Vitamin D deficiency is common in the general population and more common in children with chronic kidney disease. Vitamin D is very important for bone health, especially in children with chronic kidney disease. To date, several studies using different doses of vitamin D have been tried to correct vitamin D deficiency, but none has been completely successful. The investigators are comparing two different doses of vitamin D to determine which one is more effective at correcting and maintaining normal blood levels of vitamin D. The investigators hypothesize that a higher percentage of children receiving a higher dose of vitamin D will be vitamin D replete at the end of 6 months.

This study will enroll 80 children 9 to 18 years old who have chronic kidney disease (CKD) and can take pills. They will be enrolled from Chronic Renal Insufficiency Clinic, the Hemodialysis Unit, Peritoneal Dialysis Clinic and Transplant Clinic at Children's Healthcare of Atlanta.

DETAILED DESCRIPTION:
Vitamin D has a critical role in bone metabolism. In addition, there is increasing evidence that vitamin D has an important role in many other areas, including cardiovascular health, immune function, and prevention of autoimmune diseases and certain malignancies. In patients with CKD, there are a variety of abnormalities in mineral metabolism that lead to bone disease.

After the investigators obtain informed consent and assent, children will be randomly assigned to either low dose (1000 units daily) or high dose (4000 units daily) vitamin D pills (50% in each group). Participants will take vitamin D capsules every day for for 6 months. Vitamin D levels will be obtained at baseline, 3 months and 6 months. The study visits will be at the same time as routine clinic visits when the children are having blood drawn for routine care. At the end of the study, the investigators will compare the percentage of patients who have normal vitamin D levels at 6 months in the two groups. The investigators will also describe the percentage of patients who have elevated or low levels of trace elements.

The two doses of vitamin D in this study are within the dosing range recommended by the Institute of Medicine, and thus the investigators do not anticipate any adverse effects. Vitamin D toxicity could theoretically occur, and an elevated vitamin D level at 3 months would be an indication to withdraw a patient from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent/legal guardian must be willing and able to give written informed consent and the patient must be willing to give written informed assent if applicable
2. Estimated glomerular filtration rate < 60 mL/min/1.73 m2 body surface area or recipient of a kidney transplant
3. 9-21 years old
4. Able to swallow pills

Exclusion Criteria:

1. Liver failure
2. Malabsorption
3. Current calcium level >10.5 mg/dL
4. History of hypercalcemia (Ca >11 mg/dL) during the preceding 6 months
5. Current treatment with an antiepileptic drug or other medications that may affect vitamin D metabolism (e.g., phenobarbital, phenytoin, rifampicin)
6. History of hypervitaminosis D
7. Completion of a course of high dose vitamin D within the preceding 2 months

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-09-26 (Actual); Study Completion 2014-09-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adequate Vitamin D Level | Month 6
  Vitamin D sufficiency will be assessed as the percentage of participants with a vitamin D level >30 ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Greenbaum, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Childen's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Nadeem S, Tangpricha V, Ziegler TR, Rhodes JE, Leong T, Xiang Y, Greenbaum LA. Randomized trial of two maintenance doses of vitamin D in children with chronic kidney disease. Pediatr Nephrol. 2022 Feb;37(2):415-422. doi: 10.1007/s00467-021-05228-z. Epub 2021 Aug 15. PMID 34392411